CLINICAL TRIAL: NCT03605758
Title: A Comparative Study of Two Regimens of Ivermectin for the Treatment of Strongyloides Stercoralis Infection
Brief Title: Treatment of Strongyloides Infection
Acronym: TSSI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The original study PI passed away. Primary and Study Completion dates revised to reflect last participant examination date.
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-233
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Strongyloides Stercoralis Infection; Strongyloidiasis
Keywords: Ivermectin; S. stercoralis; parasite; helminth; Filariform; larvae; Baermann technique
MeSH Terms: conditions — Strongyloidiasis | interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Ivermectin on Days 1 and 2 (Active Comparator): Participants will receive 200 µg/kg of ivermectin daily for two consecutive days with breakfast.
  Interventions: Drug: Ivermectin
- Ivermectin on Days 1 and 14 (Active Comparator): Participants will receive 200 µg/kg of ivermectin on day one and day 14 with breakfast.
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Ivermectin is an anti-parasitic
  Other Names: Stromectol

SUMMARY:
The aim of this study is to evaluate the serologic response in patients with S. stercoralis infection after treatment with a regimen of two single doses of 200 µg/kg of ivermectin given 2 weeks apart versus a regimen of two single doses of 200 µg/kg of ivermectin given in two consecutive days.

DETAILED DESCRIPTION:
Patients will be randomly assigned to receive 2 single doses of ivermectin at 200 µg/kg 2 weeks apart versus ivermectin at 200 µg/kg for 2 consecutive days. Patients will be randomized 50-50 to the study groups using the date of birth and a random number table. All patients will be interviewed to obtain the medical history during the initial evaluation. Patients will be asked about demographic data on a questionnaire written in English and Spanish. Physical exams, baseline blood cell counts, serum chemistries, HTLV-1(human T-cell lymphotrophic virus) serology, an IgE (immunoglobulin E), a stool sample for O &P, and a pregnancy test will be performed as routine care all patients currently receive in our clinic.Procedures: Strongyloides serology will be performed in the parasitology laboratory of Jacobi Hospital with an in-house ELISA that uses a 31-kDA(kilodalton) recombinant protein antigen (termed NIE) derived from L3 stage of S. stercoralis and purified from E. coli BL21 containing pET30b plasmid. Once the in-house serology is performed serum will be banked, so it can be available to run in paired with samples taken during follow up visits. Blood samples will be also collected and sent to the Laboratory of Parasitic Diseases (LPD) at the NIAID- National Institutes of Health (NIH) to perform other serological techniques including the Luciferase Immunoprecipitation Systems Assay (LIPS) based on NIE and the recombinant antigen S. stercoralis immunoreactive antigen (SsIR). In addition, stools will be collected from all patients and will be fixated in SAF(sodium acetate, acetic acid and formalin), to check for Strongyloides stercoralis larvae. If possible, fresh stool will be obtained to check for larvae using the Baermann technique and an aliquot will be frozen and sent to the NIH for DNA extraction and PCR(polymerase chain reaction as).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Positive for Strongyloides serology infection (as determined by ELISA)

Exclusion Criteria:

* Severe intestinal Strongyloides infection
* Disseminated Strongyloidiasis infection
* Pregnant and breastfeeding women
* HTLV-1 co-infection
* Patients with indeterminate results on Strongyloides serology
* Patients who are immunosuppressed
* Unable to read and understand consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Coyle, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 participants consented. One participant expired before treatment, one participant was pregnant, and one participant was unable to be accounted for before treatment. As such, 48 participants were randomized into the study.
Groups:
- Ivermectin Administered on Two Consecutive Days (Days 1 and 2): Serologic response in patients with Strongyloides stercoralis infection after treatment with a regimen of two single doses of 200 μg/kg of ivermectin given on two consecutive days
- Ivermectin Administered Two Weeks Apart (Days 1 and 14): Serologic response in patients with Strongyloides stercoralis infection after treatment with a regimen of two single doses of 200 μg/kg of ivermectin given 2 weeks apart
Period: Overall Study
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14)
Started | 22 | 26
Completed | 0 | 2
Not Completed | 22 | 24
Not completed — Lost to Follow-up | 2 | 1
Not completed — Illness | 0 | 1
Not completed — Did not complete all 3 scheduled visits | 20 | 22

BASELINE CHARACTERISTICS:
Population: Baseline demographic data was available for 48 of the 51 participants who consented.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14) | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 2 | 8 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 8 | 17
  Hispanic | 10 | 15 | 25
  Other, not specified | 1 | 3 | 4
  White | 1 | 0 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Level of Strongyloides Serology as Measured by ELISA at 3-4 Months Post-treatment
Description: The level of Strongyloides serology as measured by Enzyme-linked immunosorbent assay (ELISA) indicates presence of infection. >0.3 OD (optical density) means positive for infection while <0.29 OD means negative (no infection).
Time Frame: 3-4 months post treatment
Population: Serology samples at 3-4 months post treatment were not collected/processed and therefore serology data is not available.
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Level of Strongyloides Serology as Measured by ELISA at 6-8 Months Post-treatment
Description: as for outcome 1
Time Frame: 6-8 months post treatment
Population: Serology samples at 6-8 months post treatment were not collected/processed and therefore serology data is not available.
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Level of Strongyloides Serology as Measured by ELISA at 9-12 Months Post-treatment
Description: as for outcome 1
Time Frame: 9-12 months post treatment
Population: Serology samples at 9-12 months post treatment were not collected/processed and therefore serology data is not available.
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months post-treatment
Description: Serious adverse events and Adverse Events were not assessed in participants prior to randomization. One participant died prior to randomization and was stratified into a distinct pre-randomization arm/group.
Groups:
- Participants Assessed for Events Prior to Randomization: One participant expired prior to randomization into study.
Arm/Group | Ivermectin Administered on Two Consecutive Days (Days 1 and 2) | Ivermectin Administered Two Weeks Apart (Days 1 and 14) | Participants Assessed for Events Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26 | 1/51
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/26 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes